CLINICAL TRIAL: NCT05715944
Title: Open-Label, Single-Arm, Phase 3b Study of the Incidence of Severe COVID-19 and Adverse Events Following AZD1222 COVID-19 Vaccination in Botswana Against SARS-CoV-2, AZD1222 - ESR-21-21311
Brief Title: Incidence of COVID-19 Following Vaccination in Botswana Against SARS CoV 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Botswana Harvard AIDS Institute Partnership (Other)
Collaborators: AstraZeneca (Industry); Botswana Ministry of Health (Other Government)
Responsible Party: Principal Investigator, Joseph M Makhema, Principal Investigator, Botswana Harvard AIDS Institute Partnership
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BHP150
Record Dates: First submitted 2022-11-09; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: COVID-19
Keywords: AZD 1222; ChAdOx1
MeSH Terms: conditions — COVID-19 | interventions — ChAdOx1 nCoV-19

STUDY DESIGN:
Intervention Model Description: AZD1222-00001 is a single-arm, Open-label, Phase 3b Study of the Incidence of Severe COVID 19 and Adverse Events Following AZD1222 COVID-19 Vaccination in Botswana Against SARS-CoV-2. Study participants are adults ≥ 18 years of age who have not already received a COVID-19 vaccine primary series and/or booster. Up to 50,000 participants are to be enrolled in the study. A total of 900 enrolled participants will also participate in a sub-study assessing the immunogenicity of AZD1222. These 900 participants in the sub-cohort will have additional assessments.
  Safety is assessed for the duration of the study. AEs are recorded at 4 weeks post the first, second and booster vaccination dose and quarterly; participants are contacted via text, or telephone call as part of follow up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AZD 1222 (Experimental): AZD1222 vaccine
  Dose Formulation:
  10 mM histidine, 7.5% (w/v) sucrose, 35 mM sodium chloride, 1 mM magnesium chloride, 0.1% (w/v) polysorbate 80, 0.1 mM edetate disodium, 0.5% (w/v) ethanol, at pH 6.6
  Current/Former names/alias(es):ChAdOx1 nCoV-19
  Interventions: Drug: AZD 1222

INTERVENTIONS:
Drug: AZD 1222 — Vaccine
  Other Names: ChAdOx1 nCoV-19

SUMMARY:
The AstraZeneca Study is a single-arm, open-label, interventional, Phase 3b study to determine the incidence of laboratory-confirmed COVID-19 hospitalizations, disease severity, and deaths and attributable adverse events (AEs) in participants in Botswana given 1 to 2 injections of AZD1222 eight to twelve weeks apart as primary series and/or 1 injection as booster dose. Length of follow-up will be 6 to 12 months, depending upon at which dose a participant is enrolled.

DETAILED DESCRIPTION:
The AstraZeneca Study is an Open-Label, Single-Arm, Phase 3b Study of the incidence of severe COVID-19 and adverse events following AZD1222 COVID-19 vaccination in Botswana against SARS-CoV-2. The study enrolled adult participants >18 years (previously >40 years) in Botswana and vaccinate them with 1 to 2 doses of AZD 1222, as primary series and/or 1 dose as booster.

Primary Objectives:

1. To assess the occurrence of severe COVID-19 disease among individuals vaccinated with AZD1222 by number of vaccine doses.
2. To assess AEs among individuals vaccinated with at least one dose of AZD1222.

Secondary Objectives:

1. To assess the occurrence of COVID-19 disease among individuals vaccinated with AZD1222 by number of vaccine doses by age group, co-morbidity group, the severity of disease and the time since the last dose.
2. To estimate the incidence of symptomatic SARS-CoV-2 infections in a sub-cohort of study participants among individuals vaccinated with at least one dose of AZD1222 by number of vaccine doses

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all of the following criteria apply:

Type of Participant

* Participants who have willingness and ability to comply with study requirements/procedures (if applicable, with assistance by legally authorised representative) based on the assessment of the investigator.
* Participants who have not yet received 3 doses of COVID-19 vaccine (2 as primary series and a booster dose). Persons who have received no prior vaccination are eligible to enroll at Day 0 to start a primary series. Persons who have received a single dose of COVID-19 vaccine at least 8 week prior (note that this includes persons who have received a single dose of Johnson & Johnson vaccine) are eligible to enroll at Day 70 to complete their primary series and receive a booster dose 3 months thereafter. Persons who have received a primary series of COVID-19 vaccine at least 3 months prior are eligible to enroll at Day 170 to receive a booster.
* Informed Consent
* Capable of giving signed informed consent, as described in Appendix A, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
* Note: A separate informed consent will be used for optional sample collection.
* Provision of signed and dated written ICF prior to any mandatory study specific procedures, sampling, and analyses.
* Age
* Participant must be ≥ 18years of age at the time of signing the informed consent and residing in the catchment area of select hospitals in Botswana.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

Prior/Concomitant Therapy

* Receipt of, or planned receipt of a COVID-19 vaccine booster dose, or any medications or investigational products indicated for the prevention of SARS-CoV-2 infection or treatment of COVID-19.
* Note: For study participants who become hospitalised with COVID-19, receipt of licensed treatment options and/or participation in investigational treatment studies is permitted.
* Receipt of any vaccine (licensed or investigational) other than licensed influenza vaccines within 30 days prior to and after administration of study intervention (i.e. the first, second and booster doses). Outside these periods, other routine vaccinations are permitted as clinically indicated.
* Medical Conditions
* Hypersensitivity to the active substance or to any of the excipients listed in Section 6.1.
* The participant reports being pregnant or nursing or has a positive pregnancy test at the time of enrolment or is planning on becoming pregnant within 6 months (for those enrolled at primary series dose 1) or 3 months (for those enrolled at primary series dose 2) of the first vaccination in the study.
* Additional details are described in Section 5.2.1.
* Individuals with risk factors for or reported history of thrombosis and/or thrombocytopenia.
* Clinically significant bleeding (eg, factor deficiency, coagulopathy, or platelet disorder) or prior history of significant bleeding or bruising following intramuscular injections or venepuncture.
* History of Guillain-Barré syndrome.
* Any confirmed or suspected immunosuppressive or immunodeficient state, including Asplenia.
* Severe and/or uncontrolled cardiovascular disease, respiratory disease, gastrointestinal disease, liver disease, renal disease, endocrine disorder, and neurological illness, as judged by the investigator (mild/moderate well-controlled comorbidities are allowed).
* Any other significant disease, disorder, or finding that may significantly increase the risk to the participant because of participation in the study, affect the ability of the participant to participate in the study, or impair interpretation of the study data.
* Note: The AESIs as outlined in the CSP should be considered when evaluating a participant for this Exclusion Criteria as the presence of these AESIs, especially if untreated or uncontrolled, may be a safety risk to the participant, affect the ability of the participant to participate in the study, or impair interpretation of the study data.
* Other Criteria
* Current participation in any other research studies that would interfere with the objectives of this study. The determination of whether participation in another study would be exclusionary for a given participant will be made by the investigator/designee.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10888 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Occurrence of severe COVID-19 disease among individuals vaccinated with AZD1222, | From at least 15 days after the second or booster dose up to 12 months following the first vaccination dose
  Occurrence of hospitalizations and deaths due to laboratory-confirmed SARS CoV 2 infection
Occurrence of Adverse Events among individuals vaccinated with at least one dose AZD1222 | Up to 12 months following the first vaccination dose
  Occurrence of Serious Adverse Events and Adverse Events of Special Interest up to 12 months following the first vaccination dose

SECONDARY OUTCOMES:
Occurrence of COVID-19 disease among individuals vaccinated with AZD1222 by number of vaccine doses and vaccine exposure, by age group, comorbidity group, severity of disease, and the time since the last dose | From at least 22 days after the first dose / at least 15 days after the second or booster dose, up to 12 months following the first vaccination dose,
  * Occurrence of hospitalizations and deaths due to laboratory-confirmed SARS-CoV-2 infection from at least 22 days after the first dose / at least 15 days after the second or booster dose, up to 12 months following the first vaccination dose, by age group, comorbidity group, severity of disease, number of vaccine doses, and the time since the last dose
  * Occurrence of laboratory-confirmed symptomatic infection from at least 22 days after the first dose / at least 15 days after the second or booster dose, up to 12 months following the first vaccination dose, by age group, comorbidity group, severity of disease, number of vaccine doses, and the time since the first or second dose
Incidence of symptomatic SARS-CoV-2 infections in a sub-cohort of study participants among individuals vaccinated with at least one dose of AZD1222, by number of vaccine doses, and by vaccine exposure | From at least 22 days after the first dose / at least 15 days after the second or booster dose, up to 12 months following the first vaccination dose
  • Occurrence of laboratory-confirmed symptomatic infection from at least 22 days after the first dose / at least 15 days after the second or booster dose, up to 12 months following the first vaccination dose

OTHER OUTCOMES:
Comparing the primary endpoint of incidence of severe COVID-19 cases to the incidence before vaccination using an observed versus expected method | From at least 15 days after the last dose up to 6-12 months following the first vaccination dose received as part of the study
  • Occurrence of hospitalizations and deaths in subjects vaccinated with AZD1222 vaccine as a primary COVID-19 vaccination series or booster dose due to laboratory-confirmed SARSCoV2 infection from at least 15 days after the last dose up to 6-12 months following the first vaccination dose received as part of the study, and the occurrence in 3-month and 6-month periods before the introduction of the AZD1222 vaccine
Monitoring the genetic diversity of breakthrough SARS-CoV-2 infections in a sub-cohort of study participants | Follow up of up to one year
  • Genotypic analysis of SARS-CoV-2 from swabs collected for severe COVID-19 cases and on Day 1 illness visit in infected study participants in the sub-cohort
Estimating the occurrence of SARS-CoV-2 infections in a sub-cohort of study participants | Follow up of up to one year
  • The incidence of SARS-CoV-2 infection defined by the presence of nucleocapsid antibodies occurring post-dose of study intervention
Assessing the humoral immunogenicity of AZD1222 vaccinated participants over time in a sub-cohort of study participants | Follow up of up to one year
  * Magnitude of SARS-CoV-2 specific antibody binding and neutralization titres (geometric mean titre)
  * Seroresponse rate of SARS-CoV-2 specific antibody binding and neutralization titres
Assessing cell mediated immune responses of AZD1222 vaccinated participants over time in a sub-cohort of study participants | Follow up of up to one year
  • Quantification of (IFN-γ) ELISpot responses to SARS-CoV-2 S protein
Assessing additional immune responses following AZD1222 vaccine as a primary COVID-19 vaccination series or as a booster | Follow up of up to one year
  • Other exploratory assays for humoral and cellular immune responses may be performed based upon emerging safety, efficacy, and immunogenicity data

CONTACTS AND LOCATIONS:
Overall Officials: Joseph M Makhema, FRCP, Principal Investigator — Botswana Harvard AIDS Institute Partnership; Tendani Gaolathe, M.,Med, Study Director — University of Botswana, Botswana Harvard Health Partnership
Locations (1):
- Botswana Harvard Health Partnership, Gaborone, Botswana

IPD SHARING:
Plan to Share IPD: No